CLINICAL TRIAL: NCT01828671
Title: A Double-Blind, Randomized, Controlled Study to Examine the Glycemic Response of Corn and Soy Tortillas in Healthy Individuals.
Brief Title: A Study to Examine the Glycemic Response of Corn and Soy Tortillas in Healthy Individuals
Acronym: SOYT-2013
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Manitoba Pulse Growers (Other)
Responsible Party: Principal Investigator, Dr. Carla Taylor, Professor and Principal Investigator, University of Manitoba
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: SOYT-2013; BREB:2013:031 (Other: University of Manitoba Biomedical Research Ethics Board)
Record Dates: First submitted 2013-04-07; First posted 2013-04-11 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-05

CONDITIONS: Healthy
Keywords: Soy; Corn; Flour; Tortilla; Glycemic; Glucose,; glycemic index
MeSH Terms: conditions — Callosities

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- Oral Glucose Solution 296 ml (Active Comparator): Study Participants will consume oral glucose solution 296 mls. Blood will be sampled via capillary at time-point 0 (before the product is consumed), and 15, 30, 45, 60, 90 and 120 minutes after consumption to determine blood glucose concentrations using a glucometer. Per standard glycemic index testing protocols, this will be repeated at another visit.
  Interventions: Other: Corn Tortilla; Other: Low Soy Flour Corn Tortilla; Other: Moderate Soy Flour Corn Tortilla; Other: High Soy Flour Corn Tortilla
- Corn Tortilla (Active Comparator): Study Participants will consume 2 to 3.5 corn tortillas (12-15 cm in diameter each) with a total serving of 25 grams of available carbohydrate. Blood will be sampled via capillary at time-point 0 (before the product is consumed), and 15, 30, 45, 60, 90 and 120 minutes after consumption to determine blood glucose concentrations using a glucometer.
  Interventions: Other: Oral Glucose Solution 296 mls
- Low Soy Flour Corn Tortilla (Active Comparator): Study Participants will consume 2 to 3.5 tortillas (12-15 cm in diameter each) with a low amount of soy flour that is 25 grams of available carbohydrate. Blood will be sampled via capillary at time-point 0 (before the product is consumed), and 15, 30, 45, 60, 90 and 120 minutes after consumption to determine blood glucose concentrations using a glucometer.
  Interventions: Other: Oral Glucose Solution 296 mls
- Moderate Soy Flour Corn Tortilla (Active Comparator): Study Participants will consume 2 to 3.5 tortillas (12-15 cm in diameter each) with moderate amount of soy flour that has 25 grams of available carbohydrate. Blood will be sampled via capillary at time-point 0 (before the product is consumed), and 15, 30, 45, 60, 90 and 120 minutes after consumption to determine blood glucose concentrations using a glucometer.
  Interventions: Other: Oral Glucose Solution 296 mls
- High Soy Flour Corn Tortilla (Active Comparator): Study Participants will consume 2 to 3.5 tortillas (12-15 cm in diameter each) with a high amount soy flour that has 25 grams of available carbohydrate. Blood will be sampled via capillary at time-point 0 (before the product is consumed), and 15, 30, 45, 60, 90 and 120 minutes after consumption to determine blood glucose concentrations using a glucometer.
  Interventions: Other: Oral Glucose Solution 296 mls

INTERVENTIONS:
Other: Oral Glucose Solution 296 mls — Should the participant be eligible to participate, they will be scheduled for two separate study visits to assess the glycemic response of the oral glucose solution.
  Arms: Corn Tortilla; High Soy Flour Corn Tortilla; Low Soy Flour Corn Tortilla; Moderate Soy Flour Corn Tortilla
Other: Corn Tortilla — Should the participant be eligible to participate, they will be scheduled for a study visit to assess the glycemic response of the corn tortillas.
  Arms: Oral Glucose Solution 296 ml
Other: Low Soy Flour Corn Tortilla — Should the participant be eligible to participate, they will be scheduled for a single study visit to assess the glycemic response of corn tortillas with a low amount of soy flour.
  Arms: Oral Glucose Solution 296 ml
Other: Moderate Soy Flour Corn Tortilla — Should the participant be eligible to participate, they will be scheduled for a single study visit to assess the glycemic response of corn tortillas with a moderate amount of soy flour.
  Arms: Oral Glucose Solution 296 ml
Other: High Soy Flour Corn Tortilla — Should the participant be eligible to participate, they will be scheduled for a single study visit to assess the glycemic response of corn tortillas with a high amount of soy flour.
  Arms: Oral Glucose Solution 296 ml

SUMMARY:
Tortillas are a staple food in several cultures and are widely used to make tacos, burritos, and enchiladas. These foods are gaining a significant segment of the North American fast food and restaurant industry. From a health point of view, the addition of soy flour into corn tortillas will improve the nutritional profile of the tortillas and the presence of soy protein, dietary fibre and bioactive components has the potential to yield other health benefits. It is hypothesized that the addition of soy flour to corn tortillas will lower the glycemic index which could benefit those individuals with type 2 diabetes.

The purpose of this research is to investigate whether different levels of soy flour in corn tortillas influences the glycemic response.

DETAILED DESCRIPTION:
Soybeans are an important crop in Canada, with approximately 10% of soybean production in Manitoba. Soybeans are grown primarily for their oil. The press cake that remains following oil extraction is a good source of protein and contains bioactive ingredients such as the isoflavones. The press cake can be ground into a flour (soy flour) and used in food products. For example, a finely ground flour can be used in infant formulas as well as for meat and dairy substitutes. This research is examining other applications of soy flour in food products such as corn tortillas. Tortillas are a staple food in several cultures and are widely used to make tacos, burritos, and enchiladas. These foods are gaining a significant segment of the North American fast food and restaurant industry. From a health point of view, the addition of soy flour into corn tortillas will improve the nutritional profile of the tortillas and the presence of soy protein, dietary fibre and bioactive components has the potential to yield other health benefits. It is hypothesized that the addition of soy flour to corn tortillas will lower the glycemic index. The glycemic index describes the potential of a food to increase blood glucose post-prandially in relation to the same amount of available carbohydrate in a glucose solution. Consumption of low glycemic index foods helps to achieve better glycemic control in individuals with type 2 diabetes. Recent meta-analyses are reporting that consumption of high glycemic index foods is associated with higher risk of coronary heart disease and breast cancer in women.

The purpose of this research is to investigate whether different levels of soy flour in corn tortillas influences the glycemic response. This information will form the basis of developing food products for glycemic management in type 2 diabetes and for reducing risk of other chronic diseases.

This single site, double-blind, randomized, controlled study designed to examine the glycemic response to corn and soy tortillas in healthy individuals will recruit 10 eligible volunteers into the study who will visit the research clinic on 6 separate visits for the glycemic testing. At each visit, one of the following products will be consumed: i) 296 mls (~1 cup) of oral glucose solution; ii) 296 mls (~1 cup) of oral glucose solution for a duplicate assessment as per standard glycemic index testing protocols; iii) corn tortillas; iv) corn tortillas with a low amount of soy flour; v) corn tortillas with a moderate amount of soy flour; or vi) corn tortillas made with a higher amount of soy flour.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, greater or equal to 18 and less than or equal to 40 years of age;
* Normal blood lipid profile (total cholesterol, LDL-cholesterol, HDL- cholesterol, triglycerides) and glycated hemoglobin <6%;
* Body mass index (BMI) of 20 to 30;
* Stable regime for the past 3 months if taking vitamin and mineral/dietary/herbal supplements;
* Agree not to eat soybeans (edamame) or soy-based foods, or consume soy or isoflavone supplements while participating in this study;
* Willing to comply with the protocol requirements;
* Willing to provide informed consent.

Exclusion Criteria:

* Allergies to corn or soy flour or to corn or soy products;
* Presence of a clinically diagnosed disease affecting the circulatory, respiratory, immune, skeletal, urinary, muscular, endocrine, digestive, nervous or reproductive system that requires medical treatment;
* Taking any prescribed medication (with the exception of birth control) within the last 3 months, or taking supplements which affect glycemic control within the last 3 months;
* Cigarette/cigar smoking, current or within the last 6 months;
* Current (within the last 30 days) bacterial, viral or fungal infection, or taking over-the-counter medication within the past 72 h;
* Pregnancy or lactation.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Blood glucose as measured via capillary sampling using glucometer | 0, 15, 30, 45, 60, 90 and 120 minutes
  Blood will be sampled via capillary finger prick at time-point 0, (before the product is consumed), and 15, 30, 45, 60, 90 and 120 minutes after the first bite of the tortillas or first sip of the glucose solution to determine blood glucose concentrations using a glucometer.

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taylor, PhD, Principal Investigator — University of Manitoba
Locations (1):
- St. Boniface General Hospital - Asper Clinical Research Institute, Winnipeg, Manitoba, Canada

REFERENCES:
- [Background] Brouns F, Bjorck I, Frayn KN, Gibbs AL, Lang V, Slama G, Wolever TM. Glycaemic index methodology. Nutr Res Rev. 2005 Jun;18(1):145-71. doi: 10.1079/NRR2005100. PMID 19079901
- [Result] Makelainen H, Anttila H, Sihvonen J, Hietanen RM, Tahvonen R, Salminen E, Mikola M, Sontag-Strohm T. The effect of beta-glucan on the glycemic and insulin index. Eur J Clin Nutr. 2007 Jun;61(6):779-85. doi: 10.1038/sj.ejcn.1602561. Epub 2006 Dec 6. PMID 17151593
- See also: Canadian Center for Agri-Food Research in Health and Medicine — http://www.ccarm.ca